CLINICAL TRIAL: NCT04342169
Title: Hydroxychloroquine for Outpatients With Confirmed COVID-19
Brief Title: University of Utah COVID-19 Hydrochloroquine Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam M. Spivak, MD, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00131893
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-01

CONDITIONS: Coronavirus Infection; Coronavirus; Infectious Disease
Keywords: coronavirus; COVID-19; hydrochloroquine; placebo
MeSH Terms: conditions — Coronavirus Infections; Communicable Diseases; COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Phase 2, prospective, placebo-controlled, parallel group, randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HCQ (Experimental): Participants randomized to the HCQ arm will receive HCQ 400mg po BID x 1 day, then 200mg po BID x 4 days. The drug dose (2.4 gm over 5 days) falls at the lower end of doses proposed in various international trials, but it has proven in vitro efficacy, with a ratio of lung tissue trough concentrations to the EC50 (effective concentration to suppress 50% of viral activity) of >20.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Those randomized to placebo will receive a placebo to be taken on the same schedule.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine — HCQ 400mg po BID x 1 day, then 200mg po BID x 4 days
  Arms: HCQ
Drug: Placebo oral tablet — Placebo to be taken on the same schedule as HCQ.
  Arms: Placebo

SUMMARY:
A novel coronavirus, SARS-CoV-2, is responsible for a rapidly spreading pandemic that has reached 160 countries, infecting over 500,000 individuals and killing more than 24,000 people. SARS-CoV-2 causes an acute and potentially lethal respiratory illness, known as COVID-19, that is threatening to overwhelm health care systems due to a dramatic surge in hospitalized and critically ill patients. Patients hospitalized with COVID-19 typically have been symptomatic for 5-7 days prior to admission, indicating that there is a window during which an effective intervention could significantly alter the course of illness, lessen disease spread, and alleviate the stress on hospital resources.

There is no known treatment for COVID-19, though in vitro and one poorly controlled study have identified a potential antiviral activity for HCQ. The rationale for this clinical trial is to measure the efficacy and safety of hydroxychloroquine for reducing viral load and shedding in adult outpatients with confirmed COVID-19.

DETAILED DESCRIPTION:
Background COVID-19 is pandemic with high mortality among hospitalized patients despite a benign course in the large majority of patients infected. Limited data are available from small outpatient studies and have not shown efficacy in preventing hospitalization. Hydroxychloroquine (HCQ) and chloroquine have antiviral and immune-modulating effects, but there are no data concerning their efficacy in reducing viral load and shedding in outpatients.

Evidence supporting possible efficacy for hydroxychloroquine. In cell models, chloroquine both interferes with terminal glycosylation of the ACE2 receptor (the cell surface receptor by which SARS-CoV2 enters human cells) and increases endosomal pH, which interferes (at least in vitro) with a crucial step in viral replication.1,2 HCQ is 5x more potent than chloroquine in a Vero cell model of SARS-CoV-2 infection. In independent experiments, chloroquine has confirmed in vitro activity against SARS-CoV-2. Additionally, HCQ has in vitro efficacy against SARS-CoV-1. According to news releases, an as-yet-unpublished set of case series in China (N reportedly 120) suggests the possibility of rapid viral clearance and low rates of progression to critical illness. In addition to in vitro anti-viral effects chloroquine and HCQ appear to have immune-modulatory effects, especially via suppression of release of TNF and IL6, especially in macrophages.

Evidence against efficacy for hydroxychloroquine. Chloroquine and HCQ have been promoted as extremely broad anti-infective agents for decades. The reported effects include suppression of fungi, atypical bacteria, and viruses. Other than the effects on ACE2 glycosylation, the mechanisms invoked as evidence for efficacy against SARS-CoV-2 have also been invoked for a wide range of viruses. However, when chloroquine and HCQ have been studied in humans, neither agent has demonstrated consistent efficacy in clinical trials, including in HIV, influenza, hepatitis, and Dengue. In one trial, chloroquine resulted in increased viral replication in Chikungunya virus [Roques et al, Viruses 2018 May 17;10(5)] while in another hydroxychloroquine was associated with increased HIV viral load [Paton et al, JAMA 2012 Jul 25;308(4):353]. Expert opinion advises against HCQ for MERS, another serious coronavirus. An underpowered (n=30) study of HCQ in COVID-19 recently published in China did not demonstrate any clinical benefit [Chen et al, J Zhejiang University, 2020 March 9]. The long history of clinical failure despite in vitro anti-viral activity suggests a low probability of efficacy.

Rationale for Trial There is significant publicity concerning the potential use of HCQ in this pandemic, and many patients are seeking access to this unproven therapy. The ANZICS guidelines emphasize that novel treatments should be administered within clinical trials; the Surviving Sepsis Campaign guidelines (http://bit.ly/SSCCOVID-19) also affirm the lack of evidence to support the clinical use of (hydroxy)chloroquine. WHO guidance (https://apps.who.int/iris/bitstream/handle/10665/331446/WHO-2019-nCoV-clinical-2020.4-eng.pdf) also strongly affirms that "investigational anti-COVID-19 therapeutics should be done under ethically approved, randomized, controlled trials." The evidence thus strongly favors equipoise.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥18 years, competent to provide consent
* Within 48 hours of positive nucleic acid test for SARS-CoV-2

Exclusion Criteria:

* Patient already prescribed chloroquine or hydroxychloroquine
* Allergy to hydroxychloroquine
* History of bone marrow or solid organ transplant
* Known G6PD deficiency
* Chronic hemodialysis, peritoneal dialysis, continuous renal replacement therapy or Glomerular Filtration Rate < 20ml/min/1.73m2
* Known liver disease (e.g. Child Pugh score ≥ B or AST>2 times upper limit)
* Psoriasis
* Porphyria
* Known cardiac conduction delay (QTc > 500mSec) or taking any prescription medications known to prolong QT interval
* Concomitant use of digitalis, flecainide, amiodarone, procainamide, or propafenone
* Seizure disorder
* Prisoner
* Weight < 35kg
* Inability to follow-up - no cell phone or no address or not Spanish or English speaking
* Receipt of any experimental treatment for SARS-CoV-2 (off-label, compassionate use, or trial related) within the 30 days prior to the time of the screening evaluation
* Patient or another member of patient's household has been already enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Spivak, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment in this trial is synonymous with treatment assignment/randomization.
Groups:
- Hydroxychloroquine: Participants randomized to the HCQ arm will receive HCQ 400mg po BID x 1 day, then 200mg po BID x 4 days. The drug dose (2.4 gm over 5 days) falls at the lower end of doses proposed in various international trials, but it has proven in vitro efficacy, with a ratio of lung tissue trough concentrations to the EC50 (effective concentration to suppress 50% of viral activity) of >20.
  Hydroxychloroquine: HCQ 400mg po BID x 1 day, then 200mg po BID x 4 days
Period: Overall Study
Arm/Group | Hydroxychloroquine | Placebo
Started | 185 | 183
Completed | 89 | 89
Not Completed | 96 | 94

BASELINE CHARACTERISTICS:
Population: Randomized participants. *one person who was erroneously administered study treatment before consenting/randomization due to a participant mix up, so although this individual will be omitted from the study's ITT-based analysis they will be included in the safety analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Placebo | Total
Number analyzed (Participants) | 185 | 182 | 367
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 165 | 164 | 329
  >=65 years | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (14.70) | 41.8 (14.40) | 41.9 (14.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 86 | 176
  Male | 95 | 96 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79 | 79 | 158
  Not Hispanic or Latino | 84 | 87 | 171
  Unknown or Not Reported | 22 | 16 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 2 | 2
  White | 86 | 80 | 166
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 96 | 96 | 192
Region of Enrollment [Number; unit: participants]
  United States | 185 | 182 | 367

OUTCOME MEASURES:

1. Primary Outcome: Duration of Viral Shedding
Description: Duration of viral shedding, as defined by time from randomization to the first of two consecutive negative swabs, measured on days 1 - 14.
Time Frame: Days
Population: Those randomized with swabs collected
Measure: Mean (Standard Error); unit: Days
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 158 | 162
Days | 9.532447 (0.3707) | 10.39556 (0.3466)

2. Secondary Outcome: Duration of COVID-19-attributable Symptoms
Description: Duration of COVID-19 symptoms (through DayA15):
  this is an integer-valued outcome which is defined as date of first asymptomatic date through the start date.
  To determine the end date, first each symptom assessment from baseline through DayA15, inclusive, will be classified as symptomatic, asymptomatic, or unknown.
  A symptomatic day is one in which at least one of the core symptoms is observed to exceed the permissible threshold: not experiencing for fever and chills; extremely mild for shortness of breath, diarrhea, and muscle aches; mild for cough and tiredness. If at most one symptom level is missing on a given day and all observed core symptoms' levels are at or below the permissible threshold, the day will be classified as asymptomatic. Otherwise (i.e. if at most five of the core symptoms have a reported symptom level and none of the reported symptom levels exceeded the threshold), the day will be considered unknown.
Time Frame: Days 1-15
Population: Among ITT that were symptomatic at baseline
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 154 | 154
Days | 6 [3 to 13] | 6 [3 to 10]

3. Secondary Outcome: Hospitalization
Description: Outcome is summarized by treatment received; all other summaries show treatment assigned
Time Frame: within 14 days of enrollment
Population: Hospitalization status unknown for 33 (3 Safety) Hydroxychloroquine, and 31 (5 Safety) Placebo participants
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 152 | 151
Participants | 7 | 4

4. Secondary Outcome: Number of Participants With Viral Shedding on Day 28
Description: The definition of the persistence of viral shedding on Day 28 outcome relies heavily on the Day 28 swab and is limited to those who have a test result for the Day 28 swab or who are not known to have died on or before DayR + 30 (there is a 2 day window for collecting the Day 28 swab). If the Day 28 swab result is known, the result will be used to define the outcome ("yes" if positive, "no" if negative). Otherwise, subjects with a confirmed cessation of viral shedding when considering daily swab results from DayR + 1 to DayR + 25, inclusive (with the requirement for confirmation waived if the latest available daily result in this interval is negative), and a missing Day 28 value will be assumed to be negative on Day 28; otherwise subjects hospitalized on any of the days DayR + 26{DayR + 30 with a missing Day 28 value will be assumed to be positive on Day 28; otherwise, multiple imputation will be performed.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 185 | 182
Participants | 30 | 30

5. Secondary Outcome: Adult Household Contact Viral Acquisition
Description: This outcome will be analyzed for households with at least two adults for which no other adult besides the index study subject is positive for COVID-19 at baseline and for which the index study subject is in the ITT population. This binary outcome will be at the household level and will be a "yes" if there is a positive swab by one or more adult household contacts for any of the study-administered swabs from days DayR + 1 to DayR + 14, inclusive. If there are no positive swabs but at least one negative swab, the outcome will be a "no;" otherwise it will be missing.
Time Frame: Days 1-14
Population: Eligible households are those with at least 2 adults, where no other adult besides the index subject is positive for COVID-19 at baseline, and where another adult submitted swab samples.
Measure: Count of Units; unit: households with at least two adults for
Units Other Than Participants: households with at least two adults for
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 185 | 182
Number analyzed (households with at least two adults for) | 33 | 39
households with at least two adults for | 16 | 19

ADVERSE EVENTS:
Time Frame: Randomization through Day 14 or hospitalization, whichever occurs first.
Description: We collected AEs that were 1. serious adverse events, 2. non-serious adverse events that are considered by the investigator to be related to study drug or study procedures or of uncertain relationship, and 3. adverse events that lead to permanent discontinuation of the study drug.
Arm/Group | Hydroxychloroquine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/183
Serious Adverse Events (participants affected / at risk) | 9/185 | 6/183
Other Adverse Events (participants affected / at risk) | 0/185 | 0/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=185) | Placebo (N=183)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shoulder Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Acute appendicitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Hospitalization (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Diabetic Foot Infection (Infections and infestations) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Oxygen saturation low (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT04342169/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT04342169/SAP_001.pdf